CLINICAL TRIAL: NCT06898450
Title: A Phase 1/2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of NDI-219216 in Patients With Advanced Solid Tumors With/Without Microsatellite Instability and/or Deficient Mismatch Repair
Brief Title: A Study to Assess the Safety, Tolerability, and Efficacy of NDI-219216 in Patients With Advanced Solid Tumors.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nimbus Wadjet, Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Organization: Nimbus Therapeutics (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 9216-101
Record Dates: First submitted 2025-03-10; First posted 2025-03-27 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumors Cancer; MSI-H Cancer
Keywords: Advanced Solid Tumors; Microsatellite Instability; Deficient Mismatch Repair; Werner syndrome helicase
MeSH Terms: conditions — Microsatellite Instability; Werner Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A dose escalation (Experimental): Part A Dose Escalation will involve enrolling sequential cohorts with increasing doses of NDI-219216 administered daily in repeating 28-day treatment cycles. The Dose Limiting Toxicity review period for each cohort will be 21 days for each patient enrolled, with review by a Safety Review Committee prior to escalation to the next dose level.
  Interventions: Drug: NDI-219216
- Part B Project Optimus (Experimental): Part B will enroll up to 3 cohorts of patients randomized between up to 3 dose levels determined from Part A Dose Escalation. NDI-219216 will be administered daily in repeating 28-day treatment cycles.
  Interventions: Drug: NDI-219216
- Part C Dose Expansion (Experimental): Part C will enroll 2 groups of patients with dMMR/MSI-h status and other select criteria, utilizing the optimal dose identified from Part B. NDI-219216 will be administered daily in 28-day repeating cycles.
  Interventions: Drug: NDI-219216

INTERVENTIONS:
Drug: NDI-219216 — NDI-219216 is a highly selective small molecule inhibitor of WRN helicase activity.

SUMMARY:
The goal of this clinical trial is to learn if NDI-219216 is safe for patients, and if NDI-219216 might be a possible treatment for advanced solid tumors in the later phases of the study.

The main questions it aims to answer are:

Is NDI-219216 safe and what kinds of side effects might it cause? What kind of effects does NDI-219216 have on the body? Does NDI-219216 have any impact on tumor size?

Participants will:

Take NDI-219216 every day by mouth. Visit the clinic 6 times during Cycle 1, 2 times during Cycle 2, once a month thereafter for checkups and tests while on the study, then one time for an end of treatment visit. After the End of Study, a follow up will occur but can be done on the phone.

Keep a diary of their tablet consumption and symptoms experienced.

DETAILED DESCRIPTION:
Study 9216-101 is a first-in-human (FIH), Phase 1/2, open-label, dose escalation, dose optimization, and dose expansion study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary antitumor activity of NDI-219216 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Have unresectable and/or metastatic solid tumors (with or without MSI-H/dMMR) refractory to or intolerant to previous SoC therapy or for which no SoC therapy exists
* Presence of measurable disease according to RECIST version 1.1 except for Part A (Dose Escalation)
* Adequate bone marrow / hematologic, end-organ, and cardiovascular function
* Resolution of all acute (or toxic) adverse effects of prior therapies, radiation therapy, or surgical procedures to Grade ≤ 1 (except fatigue, alopecia, and peripheral neuropathy).

Exclusion Criteria:

* Clinically significant cardiovascular disease.
* Patients with known WRN syndrome.
* Pregnancy, breastfeeding, or intention of becoming pregnant during the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2031-10 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Part A Primary Objective: Incidence of dose limiting toxicities (DLTs) | The first 21 days of Cycle 1 (Cycle 1 is 28 days).
  Assessments will include electrocardiograms (ECGs), echocardiogram, cardiac biomarker troponin I, physical examination, vital signs (including blood pressure, pulse), and evaluation of laboratory parameters (clinical chemistry, hematology, and coagulation)
Part A Primary Outcome: • Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs), according to NCI CTCAE v5.0 | From first dose of study drug until 30 days after last dose of study drug; up to approximately 11-12 months. Each Cycle is 28 days.
  Assessments will include standard electrocardiograms (ECGs), echocardiogram, cardiac biomarker troponin I, physical examination, vital signs (including blood pressure, pulse), and evaluation of laboratory parameters (clinical chemistry, hematology, and coagulation.
Part A Primary Outcome: Incidence and severity of Treatment Emergent Adverse Events (TEAEs) and Treatment Related Adverse Events (TRAEs) as assessed by the Investigator | From first dose of study drug until 30 days after last dose of study drug; up to approximately 11-12 months. Each Cycle is 28 days.
  Assessments will include standard electrocardiograms (ECGs), echocardiogram, cardiac biomarker troponin I, physical examination, vital signs (including blood pressure, pulse), and evaluation of laboratory parameters (clinical chemistry, hematology, and coagulation).
Part B Primary Objective: Overall Response Rate (ORR) per RECIST v1.1. | From start of study treatment until end of follow-up, up to approximately 18 months. Each Cycle is 28 days.
Part B Primary Outcome: Duration of Response (DOR) per RECIST v1.1 | From the time of first occurrence of a documented response until the time of documented disease progression or death from any cause, whichever occurs first; up to approximately 18 months. Each Cycle is 28 days.
Part B Primary Outcome: Incidence and severity of AEs according to NCI CTCAE v5.0. | From first dose of study drug until 30 days after last dose of study drug; up to approximately 18 months. Each Cycle is 28 days.
  Assessments will include standard electrocardiograms (ECGs), echocardiogram, cardiac biomarker troponin I, physical examination, vital signs (including blood pressure, pulse), and evaluation of laboratory parameters (clinical chemistry, hematology, and coagulation).
Part C Primary Objective: Overall Response Rate (ORR) per RECIST v1.1. | From start of study treatment until end of follow-up, up to approximately 17 months. Each Cycle is 28 days.
Part C Primary Outcome: Duration of Response (DOR) per RECIST v1.1. | From the time of first occurrence of a documented response until the time of documented disease progression or death from any cause, whichever occurs first, up to approximately 17 months. Each Cycle is 28 days.

SECONDARY OUTCOMES:
Part A Secondary Objective: Plasma concentrations of NDI-219216 will be measured using a validated liquid chromatography-tandem mass spectrometry (LC-MS) assay. | At pre-specified timepoints on Day 1, Day 2, Day 8, Day 21, and Day 22 of Cycle 1. Cycle 1 is 28 days in length.
Part A Secondary Outcome: Maximum Plasma Concentration Observed (Cmax) of NDI-219216 | At pre-specified timepoints on Day 1, Day 2, Day 8, Day 21, and Day 22 of Cycle 1. Cycle 1 is 28 days in length.
Part A Secondary Outcome: Time of Maximum Plasma Concentration Observed (Tmax) of NDI-219216 | At pre-specified timepoints on Day 1, Day 2, Day 8, Day 21, and Day 22 of Cycle 1. Cycle 1 is 28 days in length.
Part A Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC0-last) of NDI-219216 | At pre-specified timepoints on Day 1, Day 2, Day 8, Day 21, and Day 22 of Cycle 1 from time zero to the last observable concentration. Cycle 1 is 28 days in length.
Part B Secondary Objective: Plasma concentrations of NDI-219216 will be measured using a validated liquid chromatography-tandem mass spectrometry (LC-MS) assay. | At pre-specified timepoints on Day 1, Day 2, Day 8, Day 21, and Day 22 of Cycle 1. Cycle 1 is 28 days in length.
Part B Secondary Outcome: Maximum Plasma Concentration Observed (Cmax) of NDI-219216 | At pre-specified timepoints on Day 1, Day 2, Day 8, Day 21, and Day 22 of Cycle 1. Cycle 1 is 28 days in length.
Part B Secondary Outcome: Time of Maximum Plasma Concentration Observed (Tmax) of NDI-219216 | At pre-specified timepoints on Day 1, Day 2, Day 8, Day 21, and Day 22 of Cycle 1. Cycle 1 is 28 days in length.
Part B Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC0-last) of NDI-219216 | At pre-specified timepoints on Day 1, Day 2, Day 8, Day 21, and Day 22 of Cycle 1 from time zero to the last observable concentration. Cycle 1 is 28 days in length.
Part C Secondary Objective: Incidence and severity of AEs according to NCI CTCAE v5.0. | From first dose of study drug until 30 days after last dose of study drug; up to approximately 17 months. Each Cycle is 28 days.
  Assessments will include standard electrocardiograms (ECGs), echocardiogram, cardiac biomarker troponin I, physical examination, vital signs (including blood pressure, pulse), and evaluation of laboratory parameters (clinical chemistry, hematology, and coagulation).
Part C Secondary Objective: Plasma concentrations of NDI-219216 will be measured using a validated liquid chromatography-tandem mass spectrometry (LC-MS) assay. | At pre-specified timepoints on Day 1, Day 2, Day 8, Day 21, and Day 22 of Cycle 1. Cycle 1 is 28 days in length.
Part C Secondary Objective: Maximum Plasma Concentration Observed (Cmax) of NDI-219216 | At pre-specified timepoints on Day 1, Day 2, Day 8, Day 21, and Day 22 of Cycle 1. Cycle 1 is 28 days in length.
Part C Secondary Outcome: Time of Maximum Plasma Concentration Observed (Tmax) of NDI-219216 | At pre-specified timepoints on Day 1, Day 2, Day 8, Day 21, and Day 22 of Cycle 1. Cycle 1 is 28 days in length.
Part C Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC0-last) of NDI-219216 | At pre-specified timepoints on Day 1, Day 2, Day 8, Day 21, and Day 22 of Cycle 1. Cycle 1 is 28 days in length.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Scheuber, MD, PhD, Study Director — Nimbus Therapeutics, Inc.
Locations (24):
- United States (10):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Chicago Medicine, Chicago, Illinois
  - University of Louisville James Graham Brown Cancer Center, Louisville, Kentucky
  - Cayuga Cancer Center, Ithaca, New York
  - Atrium Health Levine Cancer Institute, Charlotte, North Carolina
  - Taylor Cancer Research Center, Maumee, Ohio
  - Brown University Health, Providence, Rhode Island
  - Prisma Health Cancer Institute - Multidisciplinary Center, Greenville, South Carolina
  - University of Virginia Emily Couric Clinical Cancer Center, Charlottesville, Virginia
  - Virginia Cancer Specialists, P.C. - Fairfax, Fairfax, Virginia
- Australia (2):
  - Liverpool Hospital, Liverpool, New South Wales
  - Southern Oncology Clinical Research Unit, Bedford Park, South Australia
- Canada (3):
  - BC Cancer Center, Kelowna, British Columbia
  - Princess Margaret Cancer Center, Toronto, Ontario
  - McGill University Health Centre (MUHC), Montreal, Quebec
- France (2):
  - Hôpital Saint-Antoine - Assistance Publique-Hopitaux de Paris (AP-HP), Paris
  - Centre Hospitalier Universitaire (CHU) de Poitiers, Poitiers
- START Dublin, Dublin, Ireland
- START Lisbon, Lisbon, Portugal
- Spain (2):
  - START Barcelona, Barcelona
  - Hospital Clinico San Carlos, Madrid
- United Kingdom (3):
  - Beatson Clinical Research Facility, Glasgow
  - Sarah Cannon Research Institute UK, London
  - The Christie NHS Foundation Trust UK, Manchester

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.